CLINICAL TRIAL: NCT06512506
Title: Prospective Cohort Study of Arthroscopic Treatment of Hip Dysplasia
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2022046
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-intervention — non-intervention

SUMMARY:
On the basis of the database established in the previous stage, a cohort analysis was conducted on patients with BDDH complicated by hip arthroscopy for minimally invasive treatment of glenoid and lip injury, according to which the indications of minimally invasive surgery for BDDH patients were optimized and surgical measures were improved. Achieve accurate and rapid repair, rehabilitation and functional recovery, serve national fitness, and treat people's injuries

DETAILED DESCRIPTION:
Based on the work of the previous research group, we prospective constructed a bidirectional cohort of patients with critical hip dysplasia, and summarized the influencing factors for the surgical prognosis of patients with BDDH, so as to continuously optimize patient selection. On this basis, the cohort size was extended to analyze the difference in efficacy between arthroscopic glenolabial repair and glenolabial repair combined with soft tissue enhancement, and further improve the minimally invasive surgery to promote the efficacy of minimally invasive surgery in BDDH patients

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of borderline hip dysplasia with glenolabial injury.

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of borderline hip dysplasia with glenolabial injury. (For example, there are no clinical symptoms of simple critical hip dysplasia, and hip pain may occur when combined with glenolabial injury
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Improved Harris hip score | Preoperative, 24 months after surgery
  It is suitable for the evaluation of therapeutic effect of various hip diseases. The Harris score includes pain, function, deformity and range of motion. The lower the improved Harris score, the worse the postoperative effect.
PRO rating | Preoperative, 24 months after surgery
  Based on Patient-Reported Outcome (PRO) : Questionnaires were completed through face-to-face or telephone interviews. Patients' symptoms, function (activity restriction), pain score, quality of life and time to return to activity were evaluated comprehensively. The lower the PRO score, the worse the postoperative effect.
Cartilage damage outerbridge grading | Preoperative, 24 months after surgery
  The patient underwent hip joint MR Examination at 12 months post-operative follow-up with T2 weighted intrachondral defect and high signal

CONTACTS AND LOCATIONS:
Overall Officials: Jianquan J Wang, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital Medicial Science Research Ethics Committee, Beijing, China

IPD SHARING:
Plan to Share IPD: No